CLINICAL TRIAL: NCT04136522
Title: A Prospective Randomized Study of the Usefulness of the Artery First Approach in Pancreatic Cancer With Pancreaticoduodenectomy
Brief Title: Usefulness of the Artery First Approach in Pancreatic Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Song Cheol Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMATME
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Pancreatic Cancer, Adult; Margin, Tumor-Free; Surgery Site Fistula; Recurrence Tumor
MeSH Terms: conditions — Pancreatic cancer, adult; Margins of Excision; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional (Active Comparator): The patients who included this group will undergo conventional pancreaticoduodenectomy (PD) or pylorus preserving pancreaticoduodenectomy (PPPD). We will identify and isolate superior mesenteric vein (SMV) before pancreatic resection. The surgeon will dissect tissue around superior mesenteric artery (SMA) and uncinate process of pancreas along the SMA.
  Interventions: Procedure: conventional pancreaticoduodenectomy
- total mesopancreas excision with arterial first approach (Experimental): The patients who included this group will undergo PD or PPPD including total pancreatic mesopancreas excision and superior mesenteric artery approach. Before pancreatic transection, the surgeon will isolate superior mesenteric vein (SMV) and superior mesenteric artery (SMA). And the surgeon will dissect nerve plexus and lymph node around SMA. inferior pancreaticoduodenal artery (IPDA) and first jejunal artery will be identified and the surgeon will ligate according to surgical margin. Anastomosis will be performed as usual manners.
  Interventions: Procedure: total mesopancreas excision including superior mesenteric artery first approach

INTERVENTIONS:
Procedure: conventional pancreaticoduodenectomy — In this subgroup, the surgeon will perform pancreaticoduodenectomy without isolation of superior mesenteric artery and dissection of nerve plexus and lymph node around superior mesenteric artery.
  Arms: conventional
Procedure: total mesopancreas excision including superior mesenteric artery first approach — In this subgroup, the surgeon will identify and isolate superior mesenteric artery before pancreatic transection, they dissect soft tissues including nerve plexus and node around superior mesenteric artery.
  Arms: total mesopancreas excision with arterial first approach

SUMMARY:
This study is aimed to evaluate difference of the 2 year recurrence free survival after pancreaticoduodenectomy for pancreatic cancer between artery-first approach and conventional procedure groups.

DETAILED DESCRIPTION:
The patients will be divided into 2 groups

conventional group: The patients who included this group will undergo conventional pancreaticoduodenectomy (PD) or pylorus preserving pancreaticoduodenectomy (PPPD). We will identify and isolate superior mesenteric vein (SMV) before pancreatic resection. The surgeon will dissect tissue around superior mesenteric artery (SMA) and uncinate process of pancreas along the SMA.

Experimental group:

The patients who included this group will undergo PD or PPPD including total pancreatic mesopancreas excision and superior mesenteric artery approach. Before pancreatic transection, the surgeon will isolate superior mesenteric vein (SMV) and superior mesenteric artery (SMA). And the surgeon will dissect nerve plexus and lymph node around SMA. inferior pancreaticoduodenal artery (IPDA) and first jejunal artery will be identified and the surgeon will ligate according to surgical margin. Anastomosis will be performed as usual manners.

Postoperative manage is same in two groups. The investigators will compared 2 years recurrence free survival rate between conventional and experimental groups.

ELIGIBILITY:
Inclusion Criteria:

* Resectable pancreatic head cancer
* No systemic metastasis
* Age > 20 years
* The patients who understand informed consent and is able to agree with study

Exclusion Criteria:

* The patients who have systemic metastasis
* The patients who need neoadjuvant therapy in borderline resectable and locally advanced pancreatic cancer
* Those with active or uncontrolled infections
* Those with severe psychiatric / neurological disorders
* Alcohol or other drug addicts
* Patients with moderate or severe comorbidities who are thought to have an impact on quality of life or nutritional status (cirrhosis, chronic kidney failure, heart failure, etc.)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
2 years recurrence free survival | 2 years after surgery
  locoregional or systemic tumor recurrence after surgery within 2 years

SECONDARY OUTCOMES:
R0 resection | 7-10 days after surgery
  Microscopic tumor clearance after surgery in pathologic result
Recurrence pattern | 2 years after surgery
  locoregional recurrence: around SMA, celiac axis, remnant pancreas, systemic recurrence: liver, lung, bone

CONTACTS AND LOCATIONS:
Overall Officials: Song-Cheol Kim, MD.PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No